CLINICAL TRIAL: NCT03480009
Title: Dextromethorphan as a Novel Non-opioid Adjunctive Agent for Pain Control in Medication Abortion: a Randomized Controlled Trial
Brief Title: Dextromethorphan as a Novel Non-opioid Adjunctive Agent for Pain Control in Medication Abortion
Acronym: DexMab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Study Investigator-Sponsor (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor-Investigator, Study Investigator-Sponsor, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19020221
Record Dates: First submitted 2018-02-15; First posted 2018-03-27 (Actual); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Abortion in First Trimester
Keywords: medication abortion; dextromethorphan; pain control
MeSH Terms: conditions — Agnosia | interventions — Dextromethorphan; Acetylcysteine; microcrystalline cellulose; Cellulose; Oxycodone; oxycodone-acetaminophen; Aspirin-oxycodone hydrochloride-oxycodone terephthalate combination

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dextromethorphan, opted for narcotic prescription (Experimental): Dextromethorphan hydrobromide and patient opts for narcotics (oxycodone or other standard narcotics)
  Interventions: Drug: Dextromethorphan Hydrobromide; Drug: Oxycodone
- Placebo, opted for narcotic prescription (Placebo Comparator): Avicel PH101 (Microcrystalline Cellulose NF) and patient opts for narcotics (oxycodone or other standard narcotics)
  Interventions: Drug: Avicel PH101 (Microcrystalline Cellulose NF) for Compounding; Drug: Oxycodone
- Dextromethorphan, declined narcotic prescription (Experimental): Dextromethorphan hydrobromide and patient declines narcotic
  Interventions: Drug: Dextromethorphan Hydrobromide
- Placebo, declined narcotic prescription (Placebo Comparator): Avicel PH101 (Microcrystalline Cellulose NF) for Compounding and patient declines narcotic
  Interventions: Drug: Avicel PH101 (Microcrystalline Cellulose NF) for Compounding

INTERVENTIONS:
Drug: Dextromethorphan Hydrobromide — Dextromethorphan capsule
  Other Names: Robitussin, Delsym
  Arms: Dextromethorphan, declined narcotic prescription; Dextromethorphan, opted for narcotic prescription
Drug: Avicel PH101 (Microcrystalline Cellulose NF) for Compounding — Placebo capsule
  Other Names: Avicel
  Arms: Placebo, declined narcotic prescription; Placebo, opted for narcotic prescription
Drug: Oxycodone — Participants may opt for the narcotic receiving arms of the study, before being randomized to dextromethorphan/placebo.
  Other Names: Tylox, Percodan, OxyContin
  Arms: Dextromethorphan, opted for narcotic prescription; Placebo, opted for narcotic prescription

SUMMARY:
This study evaluates dextromethorphan as a non-opioid adjunctive medication for pain control during medication abortion. This is double-blinded, four-arm randomized controlled trial enrolling 156 women over a period of 9-12 months: Receiving narcotics+dextromethorphan, narcotics and placebo (microcrystalline cellulose), no narcotics and dextromethorphan and no narcotics and placebo (microcrystalline cellulose).

DETAILED DESCRIPTION:
Medication abortion using mifepristone and misoprostol is common, accounting for nearly one-third of abortions in the United States in 2014. Although women generally tolerate medical abortion well, pain and bleeding are common and expected side effects. Up to a quarter of women rate their pain as severe during their procedure. Pain management for medical abortion is challenging given that the most acute pain occurs at home rather than under the supervision of medical professionals. Currently there is insufficient evidence to recommend an optimal regimen for pain control in medication abortion and there are concerns surrounding narcotic prescribing and the opiate abuse epidemic. This is a four-arm, prospective, double-blind, randomized controlled trial comparing dextromethorphan administration in conjunction with the current standard regimen (NSAIDs and narcotic medication by request- commonly oxycodone or codeine) to the standard regimen alone. Pain will be evaluated by analgesia usage and self-reported pain scores. Investigators will also investigate factors influencing pain and subjective components of the patient narrative. Ideally, a non-opioid adjunct to NSAIDs or narcotics could be used to control pain and significantly curtail or avoid opioid use. Investigators seek to test the efficacy and safety of dextromethorphan as a non-narcotic analgesic for medication abortion.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over
* Willing to give voluntary consent
* English-speaking
* Eligible for medication abortion per Planned Parenthood of Western Pennsylvania protocol
* Self-reported reliable cellular phone access for the duration of study participation
* Able to receive and reply to a "test" text at time of consent
* Willing to comply with the study protocol

Exclusion Criteria:

* Use of selective serotonin reuptake inhibitors or monoamine oxidase inhibitors due to risk of Serotonin Syndrome
* Allergy to any component of the medication abortion regimen or study drug
* Has any other condition that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, complicate the interpretation of the study outcome data, or otherwise interfere with achieving the study objectives
* Anticipated use of dextromethorphan during study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be pregnant to participate
Enrollment: 156 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD MPH, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Center for Family Planning Research, Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Planned Parenthood of Western Pennsylvania, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Penney G. Treatment of pain during medical abortion. Contraception. 2006 Jul;74(1):45-7. doi: 10.1016/j.contraception.2006.03.002. Epub 2006 May 6. PMID 16781260
- [Background] Weinbroum AA, Rudick V, Paret G, Ben-Abraham R. The role of dextromethorphan in pain control. Can J Anaesth. 2000 Jun;47(6):585-96. doi: 10.1007/BF03018952. PMID 10875724
- [Background] Ilkjaer S, Nielsen PA, Bach LF, Wernberg M, Dahl JB. The effect of dextromethorphan, alone or in combination with ibuprofen, on postoperative pain after minor gynaecological surgery. Acta Anaesthesiol Scand. 2000 Aug;44(7):873-7. doi: 10.1034/j.1399-6576.2000.440715.x. PMID 10939702
- [Background] Christie A, Dagfinrud H, Dale O, Schulz T, Hagen KB. Collection of patient-reported outcomes;--text messages on mobile phones provide valid scores and high response rates. BMC Med Res Methodol. 2014 Apr 16;14:52. doi: 10.1186/1471-2288-14-52. PMID 24735061
- [Background] Practice bulletin no. 143: medical management of first-trimester abortion. Obstet Gynecol. 2014 Mar;123(3):676-692. doi: 10.1097/01.AOG.0000444454.67279.7d. PMID 24553166
- [Derived] Ferguson GP, Achilles SL, Meyn LA, Krajewski CM, Chappell CA, Vinekar K, Chen BA. Dextromethorphan as a novel nonopioid adjunctive agent for pain control with medication abortion: A randomized controlled trial. Contraception. 2023 Feb;118:109908. doi: 10.1016/j.contraception.2022.10.010. Epub 2022 Nov 2. PMID 36332661

RESULTS

PARTICIPANT FLOW:
Groups:
- Dextromethorphan, Opted for Narcotic Prescription: Dextromethorphan hydrobromide and patient opts for narcotics (oxycodone or other standard narcotics)
  Participants may opt for the narcotic receiving arms of the study, before being randomized to dextromethorphan/placebo.
- Placebo, Opted for Narcotic Prescription: Avicel PH101 (Microcrystalline Cellulose NF) and patient opts for narcotics (oxycodone or other standard narcotics)
  Participants may opt for the narcotic receiving arms of the study, before being randomized to dextromethorphan/placebo.
- Placebo, Declined Narcotic Prescription: Avicel PH101 (Microcrystalline Cellulose NF) and patient declines narcotic
Period: Overall Study
Arm/Group | Dextromethorphan, Opted for Narcotic Prescription | Placebo, Opted for Narcotic Prescription | Dextromethorphan, Declined Narcotic Prescription | Placebo, Declined Narcotic Prescription
Started | 62 | 62 | 16 | 16
Completed | 58 | 57 | 12 | 16
Not Completed | 4 | 5 | 4 | 0
Not completed — Lost to Follow-up | 4 | 5 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Due to unequal distribution during study conduct, the protocol was modified to recruit all participants rather than into study arms. Data were analyzed as: intervention stratified by narcotic prescription status.
Groups:
- Dextromethorphan, With Narcotic Prescription: Participants receiving dextromethorphan and a narcotic prescription
- Placebo, With Narcotic Prescription: Participants receiving placebo and a narcotic prescription
- Dextromethorphan, Declined Narcotic Prescription: Participants receiving dextromethorphan and declined a narcotic prescription
- Placebo, Declined Narcotic Prescription: Participants receiving placebo and declined a narcotic prescription
- Total: Total of all reporting groups
Arm/Group | Dextromethorphan, With Narcotic Prescription | Placebo, With Narcotic Prescription | Dextromethorphan, Declined Narcotic Prescription | Placebo, Declined Narcotic Prescription | Total
Number analyzed (Participants) | 62 | 62 | 16 | 16 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (5.4) | 25.8 (4.4) | 27.1 (5.0) | 26.1 (5.3) | 26.6 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 16 | 16 | 156
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : Non-Hispanic, Black | 19 | 16 | 2 | 1 | 38
  Race : Non-Hispanic, White | 38 | 38 | 10 | 11 | 97
  Hispanic, Black | 0 | 0 | 1 | 1 | 2
  Hispanic, White | 1 | 1 | 1 | 1 | 4
  Other | 4 | 7 | 2 | 2 | 15
Prior medication abortion [Count of Participants; unit: Participants] | 12 | 12 | 1 | 2 | 27

OUTCOME MEASURES:

1. Primary Outcome: Worst Pain Measurement Via Numeric Rating Scale (NRS-11)
Description: Self-reported pain measurement via text-messaging system during first 24 hours after misoprostol administration. The scale is from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain possible".
Time Frame: Over 24 hours starting from misoprostol administration
Population: Intention to treat population where all participants were analyzed as randomized. Missing worst pain responses were imputed as 10 being the worst pain possible.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Dextromethorphan, Opted for Narcotic Prescription: Participants receiving dextromethorphan and opted for a narcotic prescription
- Placebo, Opted for Narcotic Prescription: Participants receiving placebo and opted for a narcotic prescription
Arm/Group | Dextromethorphan, Opted for Narcotic Prescription | Placebo, Opted for Narcotic Prescription | Dextromethorphan, Declined Narcotic Prescription | Placebo, Declined Narcotic Prescription
Number analyzed (Participants) | 62 | 62 | 16 | 16
score on a scale | 8.0 [6.0 to 9.0] | 7.0 [5.0 to 9.0] | 7.5 [5.5 to 10.0] | 6.5 [4.0 to 8.0]
Statistical Analysis 1: Comparison: Dextromethorphan, Opted for Narcotic Prescription vs Placebo, Opted for Narcotic Prescription; Test type: Other; p = .20, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dextromethorphan, Declined Narcotic Prescription vs Placebo, Declined Narcotic Prescription; Test type: Other; p = .20, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Analgesic Usage During Medication Abortion
Description: Analgesic usage by study arm for women who received dextromethorphan vs. placebo as adjunct to routine pain management during medication abortion; missing data are for participants who did not take the specified pain medication.
Time Frame: Over 24 hours
Population: Missing data are for participants who did not take the specified pain medication
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Dextromethorphan, Opted for Narcotic Prescription | Placebo, Opted for Narcotic Prescription | Dextromethorphan, Declined Narcotic Prescription | Placebo, Declined Narcotic Prescription
Number analyzed (Participants) | 62 | 62 | 16 | 16
mg
  ibuprofen: number analyzed (Participants) | 21 | 30 | 7 | 13
  ibuprofen | 800 [400 to 1200] | 600 [400 to 1450] | 800 [600 to 1600] | 1000 [505 to 1400]
  9acetaminophen: number analyzed (Participants) | 13 | 9 | 16 | 3
  9acetaminophen | 1000 [825 to 2000] | 1300 [1000 to 2500] | 800 [600 to 1600] | 975 [500 to 2000]
  oxycodone: number analyzed (Participants) | 29 | 25 | 0 | 1
  oxycodone | 10 [10 to 20] | 15 [10 to 20] |  | 15 [15 to 15]
Statistical Analysis 1: Comparison: Dextromethorphan, Opted for Narcotic Prescription vs Placebo, Opted for Narcotic Prescription; Ibuprofen; Test type: Other; p = .81, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dextromethorphan, Opted for Narcotic Prescription vs Placebo, Opted for Narcotic Prescription; acetaminophen; Test type: Other; p = .24, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Dextromethorphan, Opted for Narcotic Prescription vs Placebo, Opted for Narcotic Prescription; oxycodone; Test type: Other; p = .54, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Dextromethorphan, Declined Narcotic Prescription vs Placebo, Declined Narcotic Prescription; Ibuprofen; Test type: Other; p = .61, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Dextromethorphan, Declined Narcotic Prescription vs Placebo, Declined Narcotic Prescription; Acetaminophen; Test type: Other; p = .24, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mean Pain Scores Via Numeric Rating Scale (NRS-11)
Description: Marginal mean pain scores via Numeric Rating Scale (NRS-11) over 24 hours. The scale is from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain possible".
Time Frame: Marginal mean pain scores over 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale (NRS-11)
Arm/Group | Dextromethorphan, Opted for Narcotic Prescription | Placebo, Opted for Narcotic Prescription | Dextromethorphan, Declined Narcotic Prescription | Placebo, Declined Narcotic Prescription
Number analyzed (Participants) | 62 | 62 | 16 | 16
score on a scale (NRS-11) | 2.93 (2.92) | 2.96 (2.76) | 2.70 (2.95) | 2.41 (2.88)
Statistical Analysis 1: Comparison: Dextromethorphan, Opted for Narcotic Prescription vs Placebo, Opted for Narcotic Prescription; Test type: Other; p = .99, Wald Chi Square; Wald Chi Square from mixed effects linear regression
Statistical Analysis 2: Comparison: Dextromethorphan, Declined Narcotic Prescription vs Placebo, Declined Narcotic Prescription; Test type: Other; p = .56, Wald Chi Square; P-value from Wald chi-square from mixed effects linear regression

4. Secondary Outcome: Number of Participants With Pain Control Satisfaction Via 4-pt Likert Scale
Description: Overall satisfaction with pain control, "4" being - "Very good" and "1" being "Very bad"
Time Frame: 24 hours after misoprostol administration
Population: There are missing data for 3 participants in the dextromethorphan group (1 that opted for a narcotic prescription and 2 that declined) and 3 participants in the placebo (opted for narcotic prescription group).
Measure: Count of Participants; unit: Participants
Groups:
- Dextromethorphan, Opted for Narcotic Prescription: Participants receiving dextromethorphan and opted for narcotic prescription
- Placebo, Opted for Narcotic Prescription: Participants receiving placebo and opted for narcotic prescription
- Dextromethorphan, Declined Narcotic Prescription: Participants receiving dextromethorphan and declined narcotic prescription
Arm/Group | Dextromethorphan, Opted for Narcotic Prescription | Placebo, Opted for Narcotic Prescription | Dextromethorphan, Declined Narcotic Prescription | Placebo, Declined Narcotic Prescription
Number analyzed (Participants) | 61 | 59 | 14 | 16
Participants
  Very poor | 3 | 0 | 0 | 0
  Poor | 11 | 4 | 5 | 3
  Good | 27 | 30 | 7 | 8
  Very good | 20 | 25 | 2 | 5
Statistical Analysis 1: Comparison: Dextromethorphan, Opted for Narcotic Prescription vs Placebo, Opted for Narcotic Prescription; Test type: Other; p = .07, Fisher Exact
Statistical Analysis 2: Comparison: Dextromethorphan, Declined Narcotic Prescription; Test type: Other; p = .50, Fisher Exact

ADVERSE EVENTS:
Time Frame: 3-5 days after enrollment
Description: Adverse events were collected using text messaging at multiple timepoints (at baseline, misoprostol administration, and 2, 5, 8, and 24 hours after misoprostol) and by phone call 3-5 days later
Arm/Group | Dextromethorphan, Opted for Narcotic Prescription | Placebo, Opted for Narcotic Prescription | Dextromethorphan, Declined Narcotic Prescription | Placebo, Declined Narcotic Prescription
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/62 | 0/62 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 36/62 | 28/62 | 11/16 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dextromethorphan, Opted for Narcotic Prescription (N=62) | Placebo, Opted for Narcotic Prescription (N=62) | Dextromethorphan, Declined Narcotic Prescription (N=16) | Placebo, Declined Narcotic Prescription (N=16)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dextromethorphan, Opted for Narcotic Prescription (N=62) | Placebo, Opted for Narcotic Prescription (N=62) | Dextromethorphan, Declined Narcotic Prescription (N=16) | Placebo, Declined Narcotic Prescription (N=16)
Chills (General disorders) | 10 | 10 | 5 | 5
Dizziness (Nervous system disorders) | 9 | 7 | 2 | 1
Drowsiness (Nervous system disorders) | 12 | 13 | 3 | 4
Nausea (Gastrointestinal disorders) | 28 | 23 | 10 | 8
Vomiting (Gastrointestinal disorders) | 14 | 14 | 6 | 3
Diarrhea (Gastrointestinal disorders) | 8 | 13 | 7 | 4
Headache (Nervous system disorders) | 6 | 3 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT03480009/Prot_SAP_000.pdf